CLINICAL TRIAL: NCT02575729
Title: Sonography-guided Steroid Injection for Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRPG8A0051
Record Dates: First submitted 2015-09-17; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Carpal Tunnel Syndrome(CTS)
Keywords: carpal tunnel syndrome; local steroid injection; sonography; sonography-guided
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inject betamethasone by sonography (Experimental): Use 5/8 in medical needles inject betamethasone 7mg (1ml) in distal wrist crease by sonography- guided. Entering skin with 30 degrees from the ulnar side of palmaris longus tandon. Changing direction of injection to prevent median nerve injury if patients feel numbness or pain in hand.
  Interventions: Drug: betamethasone
- Inject betamethasone directly (Active Comparator): Use 5/8 in medical needles inject betamethasone 7mg (1ml) in distal wrist crease directly. Entering skin with 30 degrees from the ulnar side of palmaris longus tandon. Changing direction of injection to prevent median nerve injury if patients feel numbness or pain in hand.
  Interventions: Drug: betamethasone

INTERVENTIONS:
Drug: betamethasone — Inject betamethasone on the wrist for patient with carpal tunnel syndrome with sonography- guided, directly.
  Other Names: glucocorticoid preparation

SUMMARY:
Purpose: To compare the outcome between sonography-guided steroid injection and direct steroid injection on carpal tunnel syndrome(CTS).

DETAILED DESCRIPTION:
Material and methods: We have enrolled 26 ideopathic carpal tunnel syndrome patients (minimal to moderate according to Padua's classification).Thirteen patients were allocated in sonography approach group( sonography-guided local wrist injection, SAG) and the 13 patients were placed in direct approach group(direct local injection without using sonography, DAG). One , 3 and 6 months later after injection, we performed the outcome measures, including Boston symptom and functional scale, QuickDASH, nerve conduction study and sonography. If the patients receive the second injections, we will follow their treatment outcome by phone regularly at 1,3 and 6 months after first injection. If the patients were referred to surgery, the failures of local injection were considered and we will stop follow up them. After performing all assessment, we will compare the outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* with >2 following symptoms :

  1. disrupt sleep result in nocturnal paresthesia.
  2. symptoms release by shaking hand.
  3. pain and paresthesia during grasping.
  4. any sensory symptom on first, 2th, 3th and partial 4th fingers.
* symptoms >1month.
* Padua's classification : minimal, mild, moderate)
* meet one of three diagnosis criteria of carpal tunnel syndrome.

Exclusion Criteria:

* any history can cause periphery nerve disease.
* affected side had fracture or paralysis.
* had accepted operation for carpal tunnel syndrome before.
* pregnant
* wrist or hand sprain, ulnar nerve disease cervical nerve root disease, multiple neuropathy or nerve anastomosis.
* Padua's classification: severe, extreme.
* ultrasonography show space occupying.
* patient taking anticoagulants.
* severe systemic disease.
* wrist's skin or wrist joint has infection.
* can't complete the 6 months' follow up.
* allergy to steroid.
* has cognition disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
QuickDASH | Change from Baseline data at 6 weeks

SECONDARY OUTCOMES:
Chinese version of Boston symptom and function scale for carpal tunnel syndrome, SS & FS | Change from Baseline data at 6 weeks
Record the neurological symptoms perceived by patient after injection according to their describtion | Change from Baseline data at 6 weeks
Semmes-Weinstein Monofilament test(SWMT) | Change from Baseline data at 6 weeks
2-Point Discrimination test on 2nd digit | Change from Baseline data at 6 weeks
Nerve conduction study done on the affected hand using Necolet Viking Quest | Change from Baseline data at 6 weeks
  We will record the latency, amplitude and conduction velocity retrieved from nerve conduction study of both motor neurons and sensory neuron
Sonography examination done with patients sitting, elbow flexion and forearm supination placing on table | Change from Baseline data at 6 weeks
  The test will done twice and will record the average data of both the cross-section area and the bowing distance of transverse ligament of wrist.

CONTACTS AND LOCATIONS:
Overall Officials: Pong Ya-Ping, MD, Study Chair — Rehabilitation

REFERENCES:
- [Background] Premoselli S, Sioli P, Grossi A, Cerri C. Neutral wrist splinting in carpal tunnel syndrome: a 3- and 6-months clinical and neurophysiologic follow-up evaluation of night-only splint therapy. Eura Medicophys. 2006 Jun;42(2):121-6. PMID 16767058
- [Background] Armstrong T, Devor W, Borschel L, Contreras R. Intracarpal steroid injection is safe and effective for short-term management of carpal tunnel syndrome. Muscle Nerve. 2004 Jan;29(1):82-8. doi: 10.1002/mus.10512. PMID 14694502
- [Background] Dammers JW, Veering MM, Vermeulen M. Injection with methylprednisolone proximal to the carpal tunnel: randomised double blind trial. BMJ. 1999 Oct 2;319(7214):884-6. doi: 10.1136/bmj.319.7214.884. PMID 10506042
- [Background] Jarvik JG, Comstock BA, Kliot M, Turner JA, Chan L, Heagerty PJ, Hollingworth W, Kerrigan CL, Deyo RA. Surgery versus non-surgical therapy for carpal tunnel syndrome: a randomised parallel-group trial. Lancet. 2009 Sep 26;374(9695):1074-81. doi: 10.1016/S0140-6736(09)61517-8. PMID 19782873
- [Background] Irvine J, Chong SL, Amirjani N, Chan KM. Double-blind randomized controlled trial of low-level laser therapy in carpal tunnel syndrome. Muscle Nerve. 2004 Aug;30(2):182-7. doi: 10.1002/mus.20095. PMID 15266633
- [Background] Oztas O, Turan B, Bora I, Karakaya MK. Ultrasound therapy effect in carpal tunnel syndrome. Arch Phys Med Rehabil. 1998 Dec;79(12):1540-4. doi: 10.1016/s0003-9993(98)90416-6. PMID 9862296
- [Background] Weintraub MI, Cole SP. A randomized controlled trial of the effects of a combination of static and dynamic magnetic fields on carpal tunnel syndrome. Pain Med. 2008 Jul-Aug;9(5):493-504. doi: 10.1111/j.1526-4637.2007.00324.x. PMID 18777606
- [Background] Breuer B, Sperber K, Wallenstein S, Kiprovski K, Calapa A, Snow B, Pappagallo M. Clinically significant placebo analgesic response in a pilot trial of botulinum B in patients with hand pain and carpal tunnel syndrome. Pain Med. 2006 Jan-Feb;7(1):16-24. doi: 10.1111/j.1526-4637.2006.00084.x. PMID 16533192
- [Background] Chang MH, Chiang HT, Lee SS, Ger LP, Lo YK. Oral drug of choice in carpal tunnel syndrome. Neurology. 1998 Aug;51(2):390-3. doi: 10.1212/wnl.51.2.390. PMID 9710008
- [Background] Hui AC, Wong SM, Wong KS, Li E, Kay R, Yung P, Hung LK, Yu LM. Oral steroid in the treatment of carpal tunnel syndrome. Ann Rheum Dis. 2001 Aug;60(8):813-4. doi: 10.1136/ard.60.8.813. No abstract available. PMID 11482310
- [Background] Wong SM, Hui AC, Tang A, Ho PC, Hung LK, Wong KS, Kay R, Li E. Local vs systemic corticosteroids in the treatment of carpal tunnel syndrome. Neurology. 2001 Jun 12;56(11):1565-7. doi: 10.1212/wnl.56.11.1565. PMID 11402116
- [Background] Piazzini DB, Aprile I, Ferrara PE, Bertolini C, Tonali P, Maggi L, Rabini A, Piantelli S, Padua L. A systematic review of conservative treatment of carpal tunnel syndrome. Clin Rehabil. 2007 Apr;21(4):299-314. doi: 10.1177/0269215507077294. PMID 17613571
- [Background] Huisstede BM, Hoogvliet P, Randsdorp MS, Glerum S, van Middelkoop M, Koes BW. Carpal tunnel syndrome. Part I: effectiveness of nonsurgical treatments--a systematic review. Arch Phys Med Rehabil. 2010 Jul;91(7):981-1004. doi: 10.1016/j.apmr.2010.03.022. PMID 20599038
- [Background] Sevim S, Dogu O, Camdeviren H, Kaleagasi H, Aral M, Arslan E, Milcan A. Long-term effectiveness of steroid injections and splinting in mild and moderate carpal tunnel syndrome. Neurol Sci. 2004 Jun;25(2):48-52. doi: 10.1007/s10072-004-0229-0. PMID 15221621
- [Background] Kasten SJ, Louis DS. Carpal tunnel syndrome: a case of median nerve injection injury and a safe and effective method for injecting the carpal tunnel. J Fam Pract. 1996 Jul;43(1):79-82. PMID 8691185
- [Background] Linskey ME, Segal R. Median nerve injury from local steroid injection in carpal tunnel syndrome. Neurosurgery. 1990 Mar;26(3):512-5. doi: 10.1097/00006123-199003000-00021. PMID 2320220
- [Background] Wang LY, Leong CP, Huang YC, Hung JW, Cheung SM, Pong YP. Best diagnostic criterion in high-resolution ultrasonography for carpal tunnel syndrome. Chang Gung Med J. 2008 Sep-Oct;31(5):469-76. PMID 19097594
- [Background] Mondelli M, Filippou G, Aretini A, Frediani B, Reale F. Ultrasonography before and after surgery in carpal tunnel syndrome and relationship with clinical and electrophysiological findings. A new outcome predictor? Scand J Rheumatol. 2008 May-Jun;37(3):219-24. doi: 10.1080/03009740801914850. PMID 18465458
- [Background] Gelberman RH, Aronson D, Weisman MH. Carpal-tunnel syndrome. Results of a prospective trial of steroid injection and splinting. J Bone Joint Surg Am. 1980 Oct;62(7):1181-4. PMID 7000789